CLINICAL TRIAL: NCT01420055
Title: A 4-month, Prospective, Open-label, Multi-center Phase IV Study to Assess Response to Fingolimod Initiation According to Coping Profile in Adult Patients With Highly Active Relapsing Remitting Multiple Sclerosis in France
Brief Title: Fingolimod -Response According to Coping - Evaluation
Acronym: GRACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720DFR03; 2011-001280-49 (EudraCT Number)
Record Dates: First submitted 2011-08-17; First posted 2011-08-19 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple sclerosis; Fingolimod; Coping; Anxiety; France; Treatment Satisfaction Questionnaire for Medication-9 items (TSQM 9); Active
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Anxiety Disorders; Motor Activity | interventions — Fingolimod Hydrochloride

ARMS (1):
- fingolimod (Experimental)
  Interventions: Drug: fingolimod

INTERVENTIONS:
Drug: fingolimod

SUMMARY:
This is a prospective, open-label, multi-center phase IV study to assess response to fingolimod initiation according to coping profile in adult patients with highly active relapsing remitting multiple sclerosis in France.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 year-old male & female with RRMS (2005 revised McDonald criteria) corresponding to fingolimod indication (in Europe) and EDSS score 0 - 5.5 inclusive

Exclusion Criteria:

* History of immune system chronic disease other than MS or known immunodeficiency syndrome; increased risk for opportunistic infections, including immunocompromised patients; severe active infections, active chronic infections; negative for varicella-zoster virus IgG antibodies; live or live attenuated vaccines;
* Active malignancies; Macular edema; Cardiac disease or medicines decreasing heart rate; severe liver impairment; lymphocyte count <800/mm3;
* Pregnant or nursing (lactating) women /child-bearing potential UNLESS they are using an effective contraceptive method;
* Hypersensitivity; participation in any clinical research study within 6 months prior to baseline; prior participation in a trial with fingolimod

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To assess the mean change in Hospital Anxiety Depression Scale (HADS) anxiety sub-score between baseline and Month 4 in RRMS fingolimod treated patient total population, and according to coping profile (task, emotion or avoidance oriented). | 4 months

SECONDARY OUTCOMES:
To assess patient Clinical Global Impression (CGI) and clinician CGI at M4 in total population, and according to coping profile. | 4 months
To evaluate the safety and tolerability of fingolimod 0.5 mg/day (especially initial cardiac effects, liver function and macular edema onset) | 4 months
To explore treatment satisfaction with fingolimod in patients with RRMS either naive (rapidly evolving severe RRMS) or who transitioned from previous treatment with Disease Modifying Therapy using the TSQM 9 and according to coping profile | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (45):
- France (45):
  - Novartis Investigative Site, Angers, France
  - Novartis Investigative Site, Agen
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Auxerre
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Bayonne
  - Novartis Investigative Site, Béziers
  - Novartis Investigative Site, Bobigny
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Calais
  - Novartis Investigative Site, Castelnau-le-Lez
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, Cherbourg
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Épinal
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Hagueneau
  - Novartis Investigative Site, La Rochelle
  - Novartis Investigative Site, La Seyne-sur-Mer
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Metz
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Orsay
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Pontoise
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Roanne
  - Novartis Investigative Site, Saint-Aubin-sur-Scie
  - Novartis Investigative Site, Saint-Jean
  - Novartis Investigative Site, Sainte-Foy-lès-Lyon
  - Novartis Investigative Site, Saumur
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Talant
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tourcoing
  - Novartis Investigative Site, Tours